CLINICAL TRIAL: NCT02436798
Title: 5-HT3 Antagonists (Antiemetics) and Cardiac Safety Using an Active Surveillance Approach
Brief Title: 5-HT3 Antagonists (Antiemetics) and Cardiac Safety
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bruce Carleton, Director, Pharmaceutical Outcomes Programme, University of British Columbia
Other Study IDs: H13-02338
Record Dates: First submitted 2015-04-01; First posted 2015-05-07 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Adverse Reaction to Other Drugs and Medicines
Keywords: QT prolongation; Genomic biomarkers
MeSH Terms: conditions — Long QT Syndrome | interventions — Ondansetron

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples will be retained for genomic analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric patients: Children <6 months to 18 years of age receiving ondansetron for management of:
  1. Post-operative nausea and vomiting
  2. Chemotherapy-induced nausea and vomiting
  Interventions: Drug: Ondansetron
- Female patients: Pregnant patients or women of a reproductive age (18-45 years) receiving ondansetron for management of:
  1. Hyperemesis gravidarum
  2. Post-operative nausea and vomiting
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — All patients will be receiving treatment with ondansetron as part of standard care.
  Other Names: Zofran

SUMMARY:
5-HT3 antagonists (ondansetron) are highly effective medications for the treatment of nausea and vomiting. However, these medications also associated with potentially severe and life-threatening cardiac adverse drug reactions (ADRs), particularly QT prolongation. Data regarding the cardiac safety and inter-individual variability in cardiac effects of ondansetron when used in vulnerable populations such as children and pregnant women are very limited. The results of this study will enable better-informed therapeutic decision-making regarding the use of ondansetron in children and pregnant women, with the overall goal to improve the safety of these commonly used antiemetic medications. Furthermore, predictive pharmacogenetic markers of severe 5-HT3 antagonist toxicity could be used to identify patients at risk of cardiac toxicity before the drug is administered.

DETAILED DESCRIPTION:
The specific objectives are to:

1. Determine and compare the cardiac safety profile of ondansetron in children, when used for prevention and management of post-operative nausea and vomiting and chemotherapy induced nausea and vomiting. Identify clinical factors including pre-existing cardiac conditions or physiological conditions that predispose to ventricular arrhythmias, concomitant cardiotoxic chemotherapy or concomitant volatile anaesthetic agents and investigate their impact on cardiac adverse effects of ondansetron.
2. Determine and compare the cardiac safety profile of ondansetron when used in pregnant women or women of a reproductive age for the treatment of hyperemesis gravidarum or post-operative nausea and vomiting. Identify clinical factors including pre-existing cardiac conditions or physiological conditions, which predispose to ventricular arrhythmias that may support implementation of risk mitigation actions.
3. Identify genetic variants associated with 5-HT3 antagonist-induced prolongation of QT interval.

ELIGIBILITY:
Inclusion Criteria:

1. Children 6 months - 18 years of age who are being treated with ondansetron for prevention and management of post-operative nausea and vomiting and chemotherapy-induced nausea and vomiting.
2. Pregnant women and women of a reproductive age (18-45 years of age) who are being treated with ondansetron for hyperemesis gravidarum or postoperative nausea and vomiting.

Exclusion Criteria:

1. Patients with congenital long QT syndrome.
2. Subjects who do not speak and understand English.

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, women of a reproductive age, and pregnant women receiving ondansetron for treatment of post-operative or chemotherapy-induced nausea and vomiting or hyperemesis gravidarum.
Sampling Method: Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2014-06; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Identify clinical and genetic variants associated with ondansetron-induced prolongation of QT interval | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Carleton, PharmD., Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada